CLINICAL TRIAL: NCT06390345
Title: Functional Improvement in OSA and COPD With a Telehealth LifeStyle and Exercise Intervention
Acronym: FOCuSEd
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1766415; TE-2022C3-30598 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Obstructive Sleep Apnea; Overweight and Obesity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOCuSEd Intervention (Active Comparator): Participants randomized to the intervention will receive an integrated telehealth-delivered intervention composed of a self-directed lifestyle program and supervised pulmonary rehabilitation.
  Interventions: Other: FOCuSEd Integrated Intervention
- Usual Care- Enhanced (Active Comparator): For participants in the "enhanced" usual care group, study staff will prompt the patient's primary care provider to refer them to existing weight loss management and pulmonary rehabilitation programs.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: FOCuSEd Integrated Intervention — Participants randomized to the intervention will receive an integrated telehealth-delivered, remote lifestyle intervention that promotes healthy eating and 150 minutes per week of moderate-intensity physical exercise. This intervention will include a "core curriculum" during the first 3 months that includes: 1) a 12-session video based program; 2) goal setting and self-monitoring using a Fitbit tracker and MyFitnessPal; 3) lifestyle coaching; and 4) three tele-pulmonary rehab sessions and an additional 60-75 minutes of gradually increasing self-directed exercise per week. At the end of 3 months, we will offer to enter a recommendation for weight loss medications to intervention participants with a BMI of ≥ 27 kg/m2. In the post-core period (months 4-12), participants will continue to have as-needed access to the lifestyle coach.
  Arms: FOCuSEd Intervention
Other: Enhanced Usual Care — Participants in the "enhanced" usual care group will be referred to MOVE! (VA's weight loss management program) and pulmonary rehabilitation in coordination with their primary care provider.
  Arms: Usual Care- Enhanced

SUMMARY:
The investigators will conduct a Type I hybrid effectiveness-implementation study to test an integrated telehealth intervention among 400 overweight and obese patients with Chronic Obstructive Pulmonary Disease (COPD) and Obstructive Sleep Apnea (OSA). The investigators will include eligible participants receiving primary care at one of five Department of Veterans Affairs (VA) medical centers and their community-based outpatient clinics. The investigators will randomize patients in a 1:1 ratio to the multi-component intervention or "enhanced" usual care, stratifying by age (≥65 vs. < 65) and site. Participants randomized to the intervention will receive an integrated, telehealth-delivered intervention composed of a self-directed lifestyle program and supervised pulmonary rehabilitation. At the end of 3 months, the investigators will offer to enter a recommendation for weight management medications on behalf of eligible intervention participants. In the post-core period (months 4-12), participants will continue to have as-needed access to the lifestyle coach. For participants randomized to the "enhanced" usual care group, study staff will prompt the patient's primary care provider to refer them to existing weight loss management and pulmonary rehabilitation programs. Follow-up will occur at virtual visits at 3 and 12 months. The primary effectiveness outcome at 1-year is quality of life measured by the SF-12 Physical Component Summary Score. Secondary effectiveness outcomes will include other measures of quality of life (including sleep related impairment), sleep disturbance, disease severity (COPD exacerbations and respiratory event index for OSA), depression, social support, weight loss and cardiovascular risk. In addition to assessing effectiveness, investigators will also conduct a concurrent implementation process evaluation using the RE-AIM framework.

ELIGIBILITY:
Inclusion Criteria:

* COPD: Defined by presence of airflow obstruction (FEV1/FVC < 0.70) on post-bronchodilator spirometry
* ≥10 pack year history of tobacco use
* Self-reported clinician diagnosis of OSA (or presence of OSA on research HSAT)
* BMI ≥ 25 kg/m2
* Symptoms of dyspnea defined by MMRC score of ≥1

Exclusion Criteria:

* Self-report of weight change >15 lbs. during prior 3 months
* Current active weight loss treatment, including: 1) research-based commercial weight loss programs (e.g., Weight Watchers, Jenny Craig, HMR, Omada, TOPS, MOVE!); 2) other weight loss or related behavioral health or wellness programs led by trained personnel (professional or lay) in the local community; 3) prescription weight loss medication within last 3 months; and scheduled bariatric surgery.
* Severe illness from any cause
* Diagnosis of bulimia or history of purging behavior
* Active enrollment in pulmonary rehabilitation
* Safety and/or adherence concerns due to severe physical or mental health issues or life expectancy < 12 months. These include but may not be limited to: unstable cardiac arrhythmias, active or recent (within one month) myocardial infarction, active or recent (within one month) COPD exacerbation, angina not well-controlled with medication, significant musculoskeletal comorbidities or physical infirmities that preclude participation in an exercise program, and the need for supplemental oxygen ≥ 5 lpm at rest or with exertion.
* Pregnant, lactating, or planning to become pregnant during the study period
* Participation in other intervention studies.
* Prisoner
* Unable to complete surveys in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
The SF-12 PCS | 1 year
  The SF-12 PCS (Short Form-12, Physical Component Score) is a health-related quality of life measure that assesses general physical functioning and well-being. SF-12 PCS scores range from 0-100 with higher scores indicating better general physical health.

SECONDARY OUTCOMES:
PROMIS Sleep-related impairment | 1 year
  The Patient Reported Outcomes Measurement Information System (PROMIS) -Sleep Related Impairment Survey. The minimum value for PROMIS Sleep Related Impairment is a T-score of 30.0, the maximum is a T-score of 80.1, and a greater value indicates greater sleep related impairment, which is a worse outcome.
PROMIS Sleep-related impairment | 3 months
  The Patient Reported Outcomes Measurement Information System (PROMIS) -Sleep Related Impairment Survey. The minimum value for PROMIS Sleep Related Impairment is a T-score of 30.0, the maximum is a T-score of 80.1, and a greater value indicates greater sleep related impairment, which is a worse outcome.
SF-12 PCS | 3 months
  The SF-12 PCS (Short Form-12, Physical Component Score) is a health-related quality of life measure that assesses general physical functioning and well-being. SF-12 PCS scores range from 0-100 with higher scores indicating better general physical health.
SF-12 MCS | 3 months
  The SF-12 MCS (Short Form-12, Mental Component Score) is a health-related quality of life measure that assesses general mental health status. SF-12 MCS scores range from 0-100 with higher scores indicating better general physical health.
SF-12 MCS | 1 year
  The SF-12 MCS (Short Form-12, Mental Component Score) is a health-related quality of life measure that assesses general mental health status. SF-12 MCS scores range from 0-100 with higher scores indicating better general physical health.
PROMIS Sleep Disturbance | 3 months
  The Patient Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance Survey. The minimum value for PROMIS Sleep Disturbance is a T-score of 28.9, the maximum is a T-score of 76.5, and a greater value indicates greater sleep disturbance, which is a worse outcome.
PROMIS Sleep Disturbance | 1 year
  The Patient Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance Survey. The minimum value for PROMIS Sleep Disturbance is a T-score of 28.9, the maximum is a T-score of 76.5, and a greater value indicates greater sleep disturbance, which is a worse outcome.
COPD exacerbation or death | 3 months
  Proportion of patients with COPD exacerbation or Death (composite outcome) [ Time Frame: 3 months after randomization ]
COPD exacerbation or death | 1 year
  Proportion of patients with COPD exacerbation or Death (composite outcome) [ Time Frame: 12 months after randomization ]
COPD Assessment Test (CAT) | 3 months
  The COPD Assessment Test (CAT) ranges from a minimum of 0 to 40, with higher score comprising a worse outcome.
COPD Assessment Test (CAT) | 1 year
  The COPD Assessment Test (CAT) ranges from a minimum of 0 to 40, with higher score comprising a worse outcome.
Weight Loss | 3 months
  Total (kg)
Weight Loss | 1 year
  Total (kg)
Clinically Significant Weight Loss | 3 months
  5% weight loss met
Clinically Significant Weight Loss | 1 year
  5% weight loss met
Cardiovascular risk score | 3 months
  Non-laboratory Framingham algorithm. The minimum value in this risk score is -2, the maximum is 32, and a higher value indicates greater risk of cardiovascular disease, which is a worse outcome.
Cardiovascular risk score | 1 year
  Non-laboratory Framingham algorithm. The minimum value in this risk score is -2, the maximum is 32, and a higher value indicates greater risk of cardiovascular disease, which is a worse outcome.
Social Support | 3 months
  Social Support for diet and exercise scales
Social Support | 1 year
  Social Support for diet and exercise scales
Depression | 3 months
  PHQ-8 Depression scale
Depression | 1 year
  PHQ-8 Depression scale
Strength and endurance | 3 months
  30 second chair stand
Strength and endurance | 1 year
  30 second chair stand
OSA Severity | 1 Year
  Home-Sleep Apnea Testing: Respiratory Event Index

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Boise VA Medical Center, Boise, Idaho
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - VA Puget Sound Health Care System, Seattle, Washington
  - Mann-Grandstaff VA Medical Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will share a de-identified data set with the Patient-Centered Outcomes Research Institute-designated repository
Supporting Information: Study Protocol, SAP, ICF
Time Frame: data will be available after 2029 for at least 6 years.